CLINICAL TRIAL: NCT03823391
Title: A Randomized, Double-Blind, Double-Dummy, Active Controlled Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Efficacy of ABBV-3373 in Subjects With Moderate to Severe Rheumatoid Arthritis
Brief Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Efficacy of ABBV-3373 in Participants With Moderate to Severe Rheumatoid Arthritis (RA)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M16-560; 2018-003053-21 (EudraCT Number)
Record Dates: First submitted 2019-01-29; First posted 2019-01-30 (Actual); Results first posted 2021-07-19 (Actual); Last update posted 2021-07-19 (Actual); Status verified 2021-06

CONDITIONS: Rheumatoid Arthritis (RA)
Keywords: Rheumatoid Arthritis (RA); ABBV-3373; Adalimumab
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — ABBV-3373; Adalimumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- ABBV-3373 Followed by Placebo (Experimental): Participants will be administered with 100 mg ABBV-3373 by intravenous infusion and placebo to adalimumab by subcutaneous injection every other week for 12 weeks. After 12 weeks, participants will receive placebo to adalimumab every other week until Week 22.
  Interventions: Drug: ABBV-3373; Drug: Placebo for adalimumab
- Adalimumab (Experimental): Participants will be administered with placebo to ABBV-3373 by intravenous infusion and 80 mg adalimumab by subcutaneous injection every other week for 12 weeks. After 12 weeks, participants will receive 80 mg adalimumab subcutaneously every other week until Week 22.
  Interventions: Drug: Placebo for ABBV-3373; Drug: Adalimumab

INTERVENTIONS:
Drug: ABBV-3373 — ABBV-3373 is administered as intravenous (IV) infusion
  Arms: ABBV-3373 Followed by Placebo
Drug: Placebo for ABBV-3373 — Placebo for ABBV-3373 is administered as IV infusion
  Arms: Adalimumab
Drug: Adalimumab — Adalimumab is administered as subcutaneous (SC) injection
  Other Names: Humira
  Arms: Adalimumab
Drug: Placebo for adalimumab — Placebo for adalimumab is administered as subcutaneous (SC) injection
  Arms: ABBV-3373 Followed by Placebo

SUMMARY:
This study will assess the safety, tolerability, and efficacy of ABBV-3373 in participants with moderately to severely active rheumatoid arthritis (RA) on background methotrexate (MTX) compared with adalimumab.

DETAILED DESCRIPTION:
This study consists of a 12-week double-blind active-controlled phase and a 12 week double-blind extension period.

In the active-controlled period of the first 12 weeks of treatment, participants are randomized to receive either ABBV-3373 100 mg intravenously (IV) every other week (EOW) or adalimumab 80 mg subcutaneously (SC) EOW according to a 2:1 ratio.

At Week 12, the administration of ABBV-3373 was to stop to assess the durability of the observed clinical effects up to 24 weeks. Participants randomized to ABBV-3373 were to receive placebo injections, whereas participants randomized into the adalimumab arm were to continue their 80 mg dosing.

ELIGIBILITY:
Inclusion Criteria:

* Participant has the clinical diagnosis of RA for > 3 months based on the 1987 American College of Rheumatology (ACR) classification criteria or 2010 ACR/European League against Rheumatism (EULAR) criteria.
* Participant meets the following disease activity criteria: >= 4 swollen joints (based on 28 joint count) and >= 4 tender joints (based on 28 joint count) at Screening and Baseline visits and disease activity score (28 joints) (DAS28) C-reactive protein (CRP) >= 3.2 at Screening.
* Participant has an incomplete response to methotrexate. Participants must have been on oral or parental MTX therapy >= 3 months and on a stable prescription of 15 to 25 mg/week (or >= 10 mg/week in participants intolerant of MTX at doses >= 15 mg/week) for >= 4 weeks prior to the first dose of study drug. Participant must be expected to be able to continue on stable dose of MTX for the duration of study participation.

Exclusion Criteria:

* Participants previously exposed to adalimumab or other anti-tumor necrosis factor (TNF) biologics.
* Participants previously exposed to non-anti-TNF biologics or targeted synthetic disease-modifying antirheumatic drugs (DMARDs) for RA, with exception of participants exposed for less than 3 months and terminated not due to lack of efficacy or intolerability.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2019-03-27 (Actual); Primary Completion 2020-04-08 (Actual); Study Completion 2020-08-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: AbbVie Inc., Study Director — AbbVie
Locations (30):
- United States (18):
  - Rheum Assoc of North Alabama /ID# 213626, Huntsville, Alabama
  - AZ Arthritis and Rheum Researc /ID# 208515, Phoenix, Arizona
  - C.V. Mehta MD, Med Corporation /ID# 213068, Hemet, California
  - Robin K. Dore MD, Inc /ID# 213045, Tustin, California
  - Inland Rheum & Osteo Med Grp /ID# 213044, Upland, California
  - Suncoast Clinical Research /ID# 213973, New Port Richey, Florida
  - Arthritis Center, Inc. /ID# 213972, Palm Harbor, Florida
  - W. Broward Rheum Assoc Inc. /ID# 211017, Tamarac, Florida
  - BayCare Medical Group, Inc. /ID# 213935, Tampa, Florida
  - Institute of Arthritis Researc /ID# 213043, Idaho Falls, Idaho
  - PRN Professional Research Network of Kansas, LLC /ID# 213046, Wichita, Kansas
  - Clinvest Research LLC /ID# 215451, Springfield, Missouri
  - Duke Early Phase Research Unit (DCRI) /ID# 213212, Durham, North Carolina
  - Paramount Medical Research Con /ID# 209042, Middleburg Heights, Ohio
  - STAT Research, Inc. /ID# 213933, Vandalia, Ohio
  - West Tennessee Research Inst /ID# 208838, Jackson, Tennessee
  - PCCR Solution /ID# 215457, Colleyville, Texas
  - Trinity Universal Research Association /ID# 209167, Plano, Texas
- Charite Research Organisation GmbH /ID# 210216, Berlin, Germany
- Hungary (4):
  - CRU Hungary Egeszsegugyi és Szolgaltato Kft. /ID# 210055, Miskolc, Borsod-Abauj Zemplen county
  - DRC Gyogyszervizsgalo Kozpont Kft. /ID# 210159, Balatonfüred, Veszprém megye
  - Budai Irgalmasrendi Korhaz /ID# 208877, Budapest
  - Debreceni Egyetem Klinikai Kozpont /ID# 210164, Debrecen
- Israel (2):
  - Rambam Health Care Campus /ID# 212747, Haifa
  - Sheba Medical Center /ID# 211339, Ramat Gan
- Academisch Medical center Amsterdam /ID# 209303, Amsterdam, North Holland, Netherlands
- Poland (2):
  - SANUS Szpital Specjalistyczny /ID# 209022, Stalowa Wola
  - Reumatika - Centrum Reumatologii NZOZ /ID# 209220, Warsaw
- Puerto Rico (2):
  - GCM Medical Group, PSC /ID# 208154, San Juan
  - Mindful Medical Research /ID# 208403, San Juan

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible data sharing regarding the clinical trials we sponsor. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information (e.g., protocols and clinical study reports), as long as the trials are not part of an ongoing or planned regulatory submission. This includes requests for clinical trial data for unlicensed products and indications.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data requests can be submitted at any time and the data will be accessible for 12 months, with possible extensions considered.
Access Criteria: Access to this clinical trial data can be requested by any qualified researchers who engage in rigorous, independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information on the process, or to submit a request, visit the following link.
URL: https://www.abbvie.com/our-science/clinical-trials/clinical-trials-data-and-information-sharing/data-and-information-sharing-with-qualified-researchers.html

REFERENCES:
- [Derived] Buttgereit F, Aelion J, Rojkovich B, Zubrzycka-Sienkiewicz A, Chen S, Yang Y, Arikan D, D'Cunha R, Pang Y, Kupper H, Radstake T, Amital H. Efficacy and Safety of ABBV-3373, a Novel Anti-Tumor Necrosis Factor Glucocorticoid Receptor Modulator Antibody-Drug Conjugate, in Adults with Moderate-to-Severe Rheumatoid Arthritis Despite Methotrexate Therapy: A Randomized, Double-Blind, Active-Controlled Proof-of-Concept Phase IIa Trial. Arthritis Rheumatol. 2023 Jun;75(6):879-889. doi: 10.1002/art.42415. Epub 2023 Apr 2. PMID 36512671
- See also: Related Info — http://www.rxabbvie.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with moderately to severely active rheumatoid arthritis (RA) on background methotrexate (MTX) were enrolled at 14 sites in the United States and Puerto Rico, Poland, Hungary, and Israel.
Pre-assignment Details: Participants were randomly assigned in a 2:1 ratio to either ABBV-3373 or adalimumab. Randomization was stratified by current use of systemic glucocorticoid (≤ 7.5 mg/d prednisone equivalent) for treatment of RA at Baseline (yes/no) and prior exposure to non-anti-tumor necrosis factor (TNF) biologics or targeted synthetic disease-modifying antirheumatic drugs (DMARDs) for less than 3 months and terminated not due to lack of efficacy or intolerance (yes/no).
Groups:
- Adalimumab: Participants were administered placebo to ABBV-3373 by intravenous (IV) infusion and 80 mg adalimumab by subcutaneous injection every other week (EOW) for 12 weeks. After 12 weeks, participants received 80 mg adalimumab subcutaneously EOW until Week 22.
- ABBV-3373 Followed by Placebo: Participants were administered 100 mg ABBV-3373 by intravenous infusion and placebo to adalimumab by subcutaneous injection every other week for 12 weeks. After 12 weeks, participants received placebo to adalimumab EOW until Week 22.
Period: Period 1: Week 1 to Week 12
Arm/Group | Adalimumab | ABBV-3373 Followed by Placebo
Started | 17 | 31
Completed | 17 | 31
Not Completed | 0 | 0
Period: Period 2: Weeks 12 to Week 24
Arm/Group | Adalimumab | ABBV-3373 Followed by Placebo
Started | 17 | 31
Completed | 15 | 30
Not Completed | 2 | 1
Not completed — Adverse Event | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS) includes all randomized participants who received at least 1 dose of the study drugs.
Groups:
- Adalimumab: Participants were administered placebo to ABBV-3373 by IV infusion and 80 mg adalimumab by subcutaneous injection EOW for 12 weeks. After 12 weeks, participants received 80 mg adalimumab subcutaneously EOW until Week 22.
- ABBV-3373 Followed by Placebo: Participants were administered 100 mg ABBV-3373 by IV infusion and placebo to adalimumab by subcutaneous injection EOW for 12 weeks. After 12 weeks, participants received placebo to adalimumab EOW until Week 22.
- Total: Total of all reporting groups
Arm/Group | Adalimumab | ABBV-3373 Followed by Placebo | Total
Number analyzed (Participants) | 17 | 31 | 48
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.0 (10.21) | 52.8 (13.14) | 53.2 (12.08)
Age, Customized [Count of Participants; unit: Participants]
  < 40 years | 0 | 5 | 5
  40 to 65 years | 13 | 21 | 34
  ≥ 65 years | 4 | 5 | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 24 | 38
  Male | 3 | 7 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 8 | 11
  Not Hispanic or Latino | 14 | 23 | 37
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 16 | 28 | 44
  Black | 1 | 2 | 3
  Other | 0 | 1 | 1
Duration of RA Symptoms [Mean (Standard Deviation); unit: years] | 5.9 (3.22) | 8.0 (8.73) | 7.2 (7.29)
Duration of RA Diagnosis [Mean (Standard Deviation); unit: years] | 3.5 (3.09) | 5.0 (6.02) | 4.5 (5.19)
Baseline Use of Systemic Glucocorticoids [Count of Participants; unit: Participants] — Randomization was stratified by current use of systemic glucocorticoid (≤ 7.5 mg/day prednisone equivalent) for treatment of rheumatoid arthritis at Baseline).
  Participants
    Yes | 5 | 11 | 16
    No | 12 | 20 | 32
Prior Exposure to Non-anti-TNF or Targeted Synthetic DMARDs [Count of Participants; unit: Participants] — Randomization was stratified by prior exposure to non-anti-TNF biologics or targeted synthetic DMARDs (< 3 months and terminated not due to lack of efficacy or intolerance).
  Participants
    Yes | 0 | 0 | 0
    No | 17 | 31 | 48
Disease Activity Score 28 C-reactive protein (DAS28[CRP]) [Mean (Standard Deviation); unit: units on a scale] — The DAS28 (CRP) is a composite index used to assess rheumatoid arthritis disease activity, calculated based on the tender joint count (out of 28 evaluated joints), swollen joint count (out of 28 evaluated joints), Patient's Global Assessment of Disease Activity (0-100 mm), and high-sensitivity C-reactive protein (hsCRP) (in mg/L). Scores on the DAS28 (CRP) range from 0.96 to approximately 10, where higher scores indicate more disease activity.
  units on a scale | 5.6 (0.71) | 5.6 (0.92) | 5.6 (0.84)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Week 12 in Disease Activity Score (DAS) 28 (C-reactive Protein [CRP])
Description: The DAS28 (CRP) is a composite index used to assess rheumatoid arthritis disease activity, calculated based on the tender joint count (out of 28 evaluated joints), swollen joint count (out of 28 evaluated joints), Patient's Global Assessment of Disease Activity (measured on a visual analog scale [VAS] from 0-100 mm), and hsCRP (in mg/L). Scores on the DAS28 (CRP) range from 0.96 to approximately 10, where higher scores indicate more disease activity. A negative change from Baseline in DAS28 (CRP) indicates improvement in disease activity.
Time Frame: Baseline and Week 12
Population: Participants in the full analysis set with non-missing Baseline and at least one post-baseline value are included in the analyses.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- Adalimumab: Participants were administered placebo to ABBV-3373 by IV infusion and 80 mg adalimumab by subcutaneous injection EOW for 12 weeks.
- ABBV-3373: Participants were administered 100 mg ABBV-3373 by IV infusion and placebo to adalimumab by subcutaneous injection EOW for 12 weeks.
Arm/Group | Adalimumab | ABBV-3373
Number analyzed (Participants) | 17 | 31
score on a scale | -2.51 (0.293) | -2.65 (0.215)
Statistical Analysis 1: Comparison: ABBV-3373; Two primary comparisons were performed between ABBV-3373 and adalimumab. The first was the comparison of ABBV-3373 to historical adalimumab reference value -2.13 based on a meta-analysis consisting of 242 subjects from 3 historical adalimumab studies in which the success criterion was 2-sided P value ≤ 0.1; Test type: Superiority; p = 0.022, Mixed-effect model repeated measurement; Analysis includes treatment, visit, stratification factors, and treatment-by-visit interaction as fixed factors and Baseline value as covariate; Least Squares (LS) Mean Difference = -0.52, 90% CI 2-sided [-0.89 to -0.15], Standard Error of Mean 0.215 — Between groups difference was a single-arm comparison of LS mean of ABBV-3373 estimated from the MMRM model above minus the historical mean of adalimumab (-2.13)
Statistical Analysis 2: Comparison: ABBV-3373; The second comparison was ABBV-3373 to adalimumab with combined in-trial and borrowed historical adalimumab data using a Bayesian historical borrowing approach in which the success criterion was posterior probability of ABBV-3373 being better than adalimumab > 95%. When borrowing 30 historical adalimumab subjects, the combined least squares mean change from Baseline was -2.29; Test type: Superiority; p = 0.899, Historical data borrowing — Posterior probability; Based on posterior distribution of means for each group, the probability of Treatment mean - Control mean < 0 given the observed data was calculated
Statistical Analysis 3: Comparison: Adalimumab vs ABBV-3373; The mean difference in change from Baseline in DAS28 (CRP) at Week 12 between ABBV-3373 and adalimumab was also estimated only based on in-study data; Test type: Superiority; p = 0.683, Mixed Effect Model Repeated Measurement; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -0.15, 90% CI 2-sided [-0.74 to 0.45], Standard Error of Mean 0.353 — Treatment difference = ABBV-3373 - Adalimumab

2. Secondary Outcome: Change From Baseline to Week 12 in Clinical Disease Activity Index (CDAI)
Description: The clinical disease activity index (CDAI) is a composite index for assessing disease activity based on the summation of the counts of tender joint count (out of 28 evaluated joints) and swollen joint count (out of 28 evaluated joints), Patient Global Assessment of Disease Activity and Physician Global Assessment of Disease Activity both measured on a VAS from 0 to 10 cm. The total CDAI score ranges from 0 to 76 with higher scores indicating higher disease activity. A negative change from Baseline indicates improvement in disease activity.
Time Frame: Baseline and Week 12
Population: Participants in the full analysis set with non-missing Baseline and at least one post-baseline value were included in the analyses.
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Adalimumab | ABBV-3373
Number analyzed (Participants) | 17 | 31
score on a scale | -26.30 (2.656) | -27.99 (1.955)
Statistical Analysis 1: Comparison: Adalimumab vs ABBV-3373; Test type: Superiority; p = 0.601, Mixed Effect Model Repeated Measurement; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -1.69, 90% CI 2-sided [-7.08 to 3.70], Standard Error of Mean 3.207 — Treatment difference = ABBV-3373 - Adalimumab

3. Secondary Outcome: Change From Baseline in Simplified Disease Activity Index (SDAI)
Description: The SDAI is the numerical sum of five outcome parameters: tender and swollen joint count (based on a 28-joint assessment), Patient Global Assessment of Disease Activity and Physician Global Assessment of Disease Activity both measured on a VAS from 0-10 cm and level of CRP (in mg/dL; normal < 1 mg/dL). The SDAI has a range from 0 to 86, with higher scores indicating higher disease activity. A negative change from Baseline indicates improvement in disease activity.
Time Frame: Baseline and Week 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Adalimumab | ABBV-3373
Number analyzed (Participants) | 17 | 31
score on a scale | -27.42 (2.659) | -28.50 (1.961)
Statistical Analysis 1: Comparison: Adalimumab vs ABBV-3373; Test type: Superiority; p = 0.737, Mixed Effect Model Repeated Measurement; [statistical method as in outcome 1, analysis 1]; LS Mean Difference = -1.08, 90% CI 2-sided [-6.47 to 4.30], Standard Error of Mean 3.205 — Treatment difference = ABBV-3373 - Adalimumab

4. Secondary Outcome: Change From Baseline to Week 12 in DAS28 (Erythrocyte Sedimentation Rate [ESR])
Description: The DAS28 (ESR) is a composite index used to assess rheumatoid arthritis disease activity, calculated based on the tender joint count (out of 28 evaluated joints), swollen joint count (out of 28 evaluated joints), Patient's Global Assessment of Disease Activity (measured on a VAS from 0-100 mm), and ESR (in mm/hr). Scores on the DAS28 (ESR) range from 0 to approximately 10, where higher scores indicate more disease activity. A negative change from Baseline indicates improvement in disease activity.
Time Frame: Baseline and Week 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Adalimumab | ABBV-3373
Number analyzed (Participants) | 17 | 31
score on a scale | -2.55 (0.344) | -2.76 (0.254)
Statistical Analysis 1: Comparison: Adalimumab vs ABBV-3373; Test type: Superiority; p = 0.612, Mixed Effect Model Repeated Measurement; Analysis included treatment, visit, stratification factors, and treatment-by-visit interaction as fixed factors and Baseline value as covariate; LS Mean Difference = -0.21, 90% CI 2-sided [-0.92 to 0.49], Standard Error of Mean 0.418 — Treatment difference = ABBV-3373 - Adalimumab

5. Secondary Outcome: Percentage of Participants Achieving Low Disease Activity (LDA) Based on DAS28 (CRP) at Week 12
Description: The DAS28 (CRP) is a composite index used to assess rheumatoid arthritis disease activity, calculated based on the tender joint count (out of 28 evaluated joints), swollen joint count (out of 28 evaluated joints), Patient's Global Assessment of Disease Activity (measured on a VAS from 0-100 mm), and hsCRP (in mg/L). Scores on the DAS28 (CRP) range from 0.96 to approximately 10, where higher scores indicate more disease activity. A DAS28 (CRP) score less than or equal to 3.2 indicates low disease activity.
Time Frame: Week 12
Population: Full analysis set; participants who prematurely discontinued from study drug prior to Week 12 or for whom DAS28 data were missing at Week 12 were considered non-responders.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Adalimumab | ABBV-3373
Number analyzed (Participants) | 17 | 31
percentage of participants | 58.8 [39.2 to 78.5] | 54.8 [40.1 to 69.5]
Statistical Analysis 1: Comparison: Adalimumab vs ABBV-3373; Test type: Superiority; p = 0.877, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusted for stratification factors; Response Rate Difference = -4.0, 90% CI 2-sided [-28.5 to 20.5] — Response rate difference = ABBV-3373 - Adalimumab

6. Secondary Outcome: Percentage of Participants With an American College of Rheumatology 50% (ACR50) Response at Week 12
Description: Participants who met the following 3 conditions for improvement from Baseline were classified as meeting the ACR50 response criteria:
  1. ≥ 50% improvement in 68-tender joint count;
  2. ≥ 50% improvement in 66-swollen joint count; and
  3. ≥ 50% improvement in at least 3 of the 5 following parameters:
     * Physician global assessment of disease activity
     * Patient global assessment of disease activity
     * Patient assessment of pain
     * Health Assessment Questionnaire - Disability Index (HAQ-DI)
     * High-sensitivity C-reactive protein (hsCRP).
Time Frame: Baseline and Week 12
Population: Full analysis set; participants who prematurely discontinued from study drug prior to Week 12 or for whom ACR data were missing at Week 12 were considered non-responders.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Adalimumab | ABBV-3373
Number analyzed (Participants) | 17 | 31
percentage of participants | 64.7 [45.6 to 83.8] | 51.6 [36.8 to 66.4]
Statistical Analysis 1: Comparison: Adalimumab vs ABBV-3373; Test type: Superiority; p = 0.426, Cochran-Mantel-Haenszel; Cochran-Mantel-Haenszel test adjusting for stratification factors; Response Rate Difference = -13.1, 90% CI 2-sided [-37.2 to 11.0] — Response rate difference = ABBV-3373 - Adalimumab

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to 70 days after last dose; the treatment duration was 12 weeks in each period.
Groups:
- Period 1: ABBV-3373: Participants received 100 mg ABBV-3373 by intravenous infusion EOW and placebo to adalimumab by subcutaneous injection EOW for 12 weeks.
- Period 1: Adalimumab: Participants received 80 mg adalimumab by subcutaneous injection EOW and placebo to ABBV-3373 by intravenous infusion EOW for 12 weeks.
- Period 2: ABBV-3773 / Placebo: Participants received placebo to adalimumab by subcutaneous injection EOW from Week 12 to Week 24.
- Period 2: Adalimumab / Adalimumab: Participants continued to receive 80 mg adalimumab by subcutaneous injection EOW from Week 12 to Week 24.
Arm/Group | Period 1: ABBV-3373 | Period 1: Adalimumab | Period 2: ABBV-3773 / Placebo | Period 2: Adalimumab / Adalimumab
All-Cause Mortality (participants affected / at risk) | 0/31 | 0/17 | 0/30 | 0/16
Serious Adverse Events (participants affected / at risk) | 4/31 | 0/17 | 0/30 | 2/16
Other Adverse Events (participants affected / at risk) | 4/31 | 12/17 | 7/30 | 12/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Period 1: ABBV-3373 (N=31) | Period 1: Adalimumab (N=17) | Period 2: ABBV-3773 / Placebo (N=30) | Period 2: Adalimumab / Adalimumab (N=16)
NON-CARDIAC CHEST PAIN (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ANAPHYLACTIC SHOCK (Immune system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
BREAST ABSCESS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
BRONCHITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PNEUMONIA (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Period 1: ABBV-3373 (N=31) | Period 1: Adalimumab (N=17) | Period 2: ABBV-3773 / Placebo (N=30) | Period 2: Adalimumab / Adalimumab (N=16)
LEUKOPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PERIORBITAL SWELLING (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
MOUTH SWELLING (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
NAUSEA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
INFUSION SITE BRUISING (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
INJECTION SITE PRURITUS (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OEDEMA PERIPHERAL (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PYREXIA (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DRUG HYPERSENSITIVITY (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
TYPE I HYPERSENSITIVITY (Immune system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
BRONCHITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
GASTROENTERITIS VIRAL (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
NASOPHARYNGITIS (Infections and infestations) | 0 (0) | 1 (1) | 3 (3) | 2 (2)
ORAL HERPES (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
SINUSITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 2 (2) | 2 (2) | 1 (1) | 1 (1)
BLOOD PRESSURE INCREASED (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
LIVER FUNCTION TEST ABNORMAL (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MYCOPLASMA TEST POSITIVE (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
RHEUMATOID ARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
HEADACHE (Nervous system disorders) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
HYPOAESTHESIA (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SCIATICA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
BRONCHIAL HYPERREACTIVITY (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PRURITUS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
HYPERTENSION (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
AbbVie requests that any investigator or institution that plans on presenting/publishing results disclosure, provide written notification of their request 60 days prior to their presentation/publication. AbbVie requests that no presentation/publication will be instituted until 12 months after a study is completed, or after the first presentation/publication whichever occurs first. A delay may be proposed of a presentation/publication if AbbVie needs to secure patent or proprietary protection.

DOCUMENTS (2):
  • Study Protocol (2020-09-04): https://cdn.clinicaltrials.gov/large-docs/91/NCT03823391/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-08): https://cdn.clinicaltrials.gov/large-docs/91/NCT03823391/SAP_001.pdf